CLINICAL TRIAL: NCT00399516
Title: The Effect of Pulse Width on the Treatment of Chronic Low Back Pain With Spinal Cord Stimulation
Brief Title: Effect of Pulse Width With Spinal Cord Stimulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCS0706
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-03

CONDITIONS: Pain; Chronic Pain; Back Pain
Keywords: Pain; Neurostimulation; Back pain; Chronic Pain
MeSH Terms: conditions — Pain; Chronic Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Precision

SUMMARY:
The primary objective of this study is to assess the effects of varying pulse width in suprathreshold dorsal column stimulation in patients with low back pain.

DETAILED DESCRIPTION:
This study will generate data which may allow Precision SCS devices to be used or programmed in such a way as to relieve pain while minimizing any uncomfortable sensations. This study will extend anecdotal reports into a prospective analysis of outcome data.

Patients invited to participate in this study will have recently been implanted with the Precision system, or will be eligible for SCS therapy and will have already selected therapy with the Advanced Bionics Precision system, independent of possible inclusion in this study.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic low back pain following spine surgery (Failed Back Surgery Syndrome), which is primarily located in the low back, with minimal lower extremity pain.
* Have been permanently implanted with a Precision spinal cord stimulation (SCS) system within 6 months, or be an appropriate candidate for SCS and for the surgical procedures required for SCS as determined by the physician and have independently selected SCS with Precision for treatment.
* Be 18 years of age or older.
* Be willing and able to comply with all study related procedures and visits.
* Be capable of reading and understanding patient information materials and giving written informed consent.

Exclusion Criteria:

* Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints.
* Have any other chronic pain condition likely to confound evaluation of study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-11; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Yearwood, MD, Principal Investigator — Comprehensive Pain and Rehabilitation
Locations (1):
- Comprehensive Pain Management and Rehabilitation, Daphne, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Cord Stimulation Programming Parameters: Spinal Cord Stimulation (SCS) treatment group programmed using a randomly assigned sequence of stimulation parameters (i.e. pulse widths)
Period: Overall Study
Arm/Group | Spinal Cord Stimulation Programming Parameters
Started | 21
Completed | 19
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Spinal Cord Stimulation Programming Parameters: Spinal Cord Stimulation (SCS) Treatment Group
Arm/Group | Spinal Cord Stimulation Programming Parameters
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Pain Severity, as Measured on the 11-point (0-10) Numerical Rating Scale (NRS)
Description: Pain severity as measured by NRS quantifies pain, where 0 is "no pain" and 10 is "worst pain imaginable"
Time Frame: Within 6 months post-implantation
Measure: Mean (Standard Deviation); unit: Percent Change in Pain Rating
Arm/Group | Spinal Cord Stimulation Programming Parameters
Number analyzed (Participants) | 19
Percent Change in Pain Rating | -56.1 (25.8)

ADVERSE EVENTS:
Arm/Group | Spinal Cord Stimulation Programming Parameters
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Cord Stimulation Programming Parameters (N=21)
Stimulation not tolerated (Nervous system disorders) | 1 (1)
Pain (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less